CLINICAL TRIAL: NCT01906814
Title: Three Cycles Versus Six Cycles of Adjuvant Chemotherapy for the Patients With High-risk Retinoblastoma After Enucleation: Prospective Randomized Control Study
Brief Title: Adjuvant Chemotherapy for High-risk Retinoblastoma After Enucleation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: yanghs20130507
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Vincristine; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 cycles chemotherapy (Experimental): Chemotherapy: vincristine 0.05 mg/kg (or 1.5 mg/m2 for children ≥ 3 years of age) on Day 1, carboplatin 18.6 mg/kg (or 560 mg/m2 for children ≥ 3 years of age) on Day 1, etoposide 5.0 mg/kg/day (or 150 mg/ m2 for children ≥ 3 years of age) on Days 1 and 2 and 2. Cycles were repeated every 21 days for three cycles.
  Interventions: Drug: 3 cycles chemotherapy
- 6 cycles chemotherapy (Active Comparator): Chemotherapy: vincristine 0.05 mg/kg (or 1.5 mg/m2 for children ≥ 3 years of age) on Day 1, carboplatin 18.6 mg/kg (or 560 mg/m2 for children ≥ 3 years of age) on Day 1, etoposide 5.0 mg/kg/day (or 150 mg/ m2 for children ≥ 3 years of age) on Days 1 and 2 and 2. Cycles were repeated every 21 days for six cycles.
  Interventions: Drug: 6 cycles chemotherapy

INTERVENTIONS:
Drug: 3 cycles chemotherapy — Chemotherapy: vincristine 0.05 mg/kg (or 1.5 mg/m2 for children ≥ 3 years of age) on Day 1, carboplatin 18.6 mg/kg (or 560 mg/m2 for children ≥ 3 years of age) on Day 1, etoposide 5.0 mg/kg/day (or 150 mg/ m2 for children ≥ 3 years of age) on Days 1 and 2 and 2. Cycles were repeated every 21 days for three cycles.
  Other Names: vincristine, carboplatin, etoposide.
  Arms: 3 cycles chemotherapy
Drug: 6 cycles chemotherapy — Chemotherapy: vincristine 0.05 mg/kg (or 1.5 mg/m2 for children ≥ 3 years of age) on Day 1, carboplatin 18.6 mg/kg (or 560 mg/m2 for children ≥ 3 years of age) on Day 1, etoposide 5.0 mg/kg/day (or 150 mg/ m2 for children ≥ 3 years of age) on Days 1 and 2 and 2. Cycles were repeated every 21 days for six cycles.
  Other Names: vincristine, carboplatin, etoposide.
  Arms: 6 cycles chemotherapy

SUMMARY:
The purpose of this study is to determine whether 3 cycles of chemotherapy(CEV) is not inferior to 6 cycles of chemotherapy(CEV) in the treatment of Stage I enucleated retinoblastoma.

DETAILED DESCRIPTION:
This study will be a phase Ⅲ open label interventional case series. Patients with unilateral Stage I enucleated retinoblastoma will be randomized to receive chemotherapy(CEV) of 3 cycles or 6 cycles every 21 days. Patients will be followed for 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Definite pathology signs of retinoblastoma, Stage I base on International Retinoblastoma Staging System.
* Received enucleation in the study eye.
* Monocular retinoblastoma.

Exclusion Criteria:

* Any previous disease in the study eye.
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals).
* History of chemical intervention for retinoblastoma in the study eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | five years
  measure the disease-free survival rate for the two groups at five years

SECONDARY OUTCOMES:
overall survival | five years
  time from randomization to death as a result of any cause at five years
safety: side effects of chemotherapy in the Treatment of Retinoblastoma | five years
  Number of participants with side effects (systemic check-up, audio acuity, ect)before each treatment, at 1,3,6,9,12,18,24,30,36,42,48,54,60 months after the treatment.
quality of life (PedsQL4.0 scale) in the Treatment of Retinoblastoma | five years
  quality of life (PedsQL4.0 scale) before each treatment, at 1,3,6,9,12,18,24,30,36,42,48,54,60 months after the treatment. PedsQL 4.0 questionnaire has two modules (reported by parents and children) with 23 items encompassing the physical domains (8 items), emotional (5 items), social (5 items) and school (5 items). A five scores scale is used, after being asked, ''How much, in the last month, your child has had problems with'' (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = is often a problem and 4 = almost always a problem). The items are reverse-score and linearly transformed to a scale from 0 to 100 (0=100, 1=75, 2=50, 3=25, 4 = 0). So high scores indicate better QoL.
economic burden due to chemotherapy | during chemotherapy (9 weeks for 3-cycle group, and 18 weeks for 6-cycle group)
  All costs, including direct cost and indirect cost, are expressed in Chinese YUAN. Direct costs include the average cost of systemic chemotherapy, operation, supportive treatment, and examination. Indirect costs include accommodation, transportation, diet, and lost income of parents.

CONTACTS AND LOCATIONS:
Overall Officials: Huasheng Yang, Doctor, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye H, Xue K, Zhang P, Chen R, Zhai X, Ling L, Xiao W, Tang L, Wang H, Mao Y, Ai S, Bi Y, Liu Q, Zou Y, Qian J, Yang H. Three vs 6 Cycles of Chemotherapy for High-Risk Retinoblastoma: A Randomized Clinical Trial. JAMA. 2024 Nov 19;332(19):1634-1641. doi: 10.1001/jama.2024.19981. PMID 39432296